CLINICAL TRIAL: NCT03692598
Title: Study of Transcatheter Tricuspid Annular Repair
Acronym: STTAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Micro Interventional Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MID-002
Record Dates: First submitted 2016-12-02; First posted 2018-10-02 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MIA Surgical (Experimental): Eligible patients will receive implantation of MIA implants deployed using the MIA, Minimally Invasive Annuloplasty Device - Surgical from an open surgical approach
  Interventions: Device: MIA, Minimally Invasive Annuloplasty Device - Surgical
- MIA Percutaneous (Experimental): Eligible patients will receive implantation of MIA implants deployed using the MIA, Minimally Invasive Annuloplasty Device - Percutaneous from a transcatheter approach
  Interventions: Device: MIA, Minimally Invasive Annuloplasty Device - Percutaneous

INTERVENTIONS:
Device: MIA, Minimally Invasive Annuloplasty Device - Surgical — Eligible patients will receive implantation of MIA implants deployed using the MIA, Minimally Invasive Annuloplasty Device from an open surgical approach
  Other Names: MIA-S
  Arms: MIA Surgical
Device: MIA, Minimally Invasive Annuloplasty Device - Percutaneous — Eligible patients will receive implantation of MIA implants deployed using the MIA, Minimally Invasive Annuloplasty Device from a percutaneous approach
  Other Names: MIA
  Arms: MIA Percutaneous

SUMMARY:
The purpose of the study is to evaluate the safety and performance of the MIA Minimally Invasive Annuloplasty Device in patients with chronic functional tricuspid regurgitation.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety and performance of the MIA Minimally Invasive Annuloplasty Device in patients with chronic functional tricuspid regurgitation. The study is a prospective, multi-center safety and performance study. Enrolled subjects will be assessed for clinical follow-up at 1 month, 6 months, and 1 year post implant procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic functional tricuspid regurgitation (FTR) with a minimum of moderate tricuspid regurgitation (2-4)
2. Age≥18 and ≤85 years old
3. New York Heart Association (NYHA) Class II, III or ambulatory IV
4. Left ventricular ejection fraction (LVEF) ≥30%
5. Undergoing cardiac surgical procedure with the planned use of cardiopulmonary bypass (surgical arm only)
6. Functional tricuspid valve regurgitation pathology with a structurally normal valve; and tricuspid valve annular diameter ≥ 40 mm (or 21 mm/m2) and ≤55 mm (or 29 mm/m2) or 2-4 + FTR
7. Patient provides written Informed Consent before any study-specific tests or procedures are performed
8. Patient is willing and able to comply with all specified study evaluations

Exclusion Criteria:

1. Pregnant or lactating female
2. Severe uncontrolled hypertension (SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg)
3. Previous tricuspid valve repair or replacement
4. Myocardial Infarction or known unstable angina within the 30-days prior to the index procedure
5. Any PCI within 30 days prior to the index procedure or planned 3 months post the index procedure
6. Life expectancy of less than 12-months
7. Severe right heart dysfunction
8. Pulmonary hypertension with PA mean 2/3 rd MAP
9. Active systemic infection
10. Pericardial infection
11. Any clinical evidence that the investigator feels would place the patient at increased risk with the deployment of the device
12. Co-morbid conditions that place the subject at an unacceptable surgical risk (e.g. severe chronic obstructive pulmonary disease, hepatic failure, cardiac disease, autoimmune disorders or conditions of severe immunosuppression)
13. Untreated coronary artery disease (CAD) requiring revascularisation unless CABG procedure is concomitant with MIA tricuspid annular repair (surgical arm only)
14. Haemodynamic instability: systolic blood pressure <90mmHg without reduction of afterload, shock, need for inotropic medication or IABP
15. Active peptic ulcer or gastrointestinal (GI) bleeding in the past 3 months
16. Cerebrovascular event within the past 6 months
17. History of mitral/tricuspid endocarditis within the last 12 months
18. Organic tricuspid disease
19. Contraindication or known allergy to device's components, aspirin, anti-coagulation therapy or contrast media that cannot be adequately premeditated
20. Known alcohol or drug abuser
21. Currently participating in the study of an investigational drug or device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Events | 30 days
  The percentage of participants with Major Adverse Events within 30 days of the procedure: death, Q-wave myocardial infarction, cardiac tamponade, cardiac surgery for failed MIA implantation, or stroke
Reduction in tricuspid regurgitation at 30 days | 30 days
  The reduction in the degree of tricuspid regurgitation compared to baseline measured post-procedure, at post-operative hospital discharge and at 1 month post-operative. Ability to reduce tricuspid regurgitation by at least 1 degree by means of quantitative echocardiographic parameters

SECONDARY OUTCOMES:
Serious Adverse Events (SAEs) and Serious Adverse Device Events (SADE) | 3 months
  The percentage of participants with Serious Adverse Events (SAEs) and Serious Adverse Device Events (SADE) within 6 months of the procedure will be compared to the literature.
Reduction in tricuspid regurgitation | 3 months
  Assessment in the degree of Tricuspid Regurgitation at 3 months compared to baseline Ability to maintain improvement in tricuspid regurgitation with respect to baseline.
Quality of Life Measurement | 3 months
  Change in quality of life questionnaire (Minnesota Living with Heart Failure Questionnaire) compared to baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kestutis Rucinskas, MD, Principal Investigator — Vilnius University Hospital, Santariskiu Klinikos
Locations (6):
- Aarhus University Hospital, Aarhus, Denmark
- Semmelweis University, Heart and Vascular Center, Budapest, Hungary
- Centre of Cardiology, Pauls Stradins Clinical University Hospital, Riga, Latvia
- Lithuania (2):
  - Lithuanian University of Health Sciences, Kaunas
  - Vilnius University Hospital Santariskiu Klinikos, Vilnius
- The Cardinal Stefan Wyszyński Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No